CLINICAL TRIAL: NCT06791889
Title: Blood DdPCR for Early Identification and Dynamic Surveillance of Pathogenic Bacteria in ICU Septic Patients: a Single-centre, Prospective, Observational Study
Status: Recruiting | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: WHUICU202409
Record Dates: First submitted 2025-01-19; First posted 2025-01-24 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Sepsis; Bloodstream Infections; Critically Ill Intensive Care Unit Patients
Keywords: ddPCR; Sepsis; ICU
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- ddPCR group

SUMMARY:
The purpose of this study is to investigate the efficacy of droplet digital PCR (ddPCR) in identifying pathogenic organisms in ICU sepsis patients, aiming to find a method that allows early identification of pathogenic organisms and dynamic surveillance in order to assess the association between pathogenic species and loads and clinical characteristics and outcomes.

DETAILED DESCRIPTION:
This is a monocentric observational study. Patients admitted to the ICU with a first diagnosis of sepsis will be dynamically monitored for nucleic acid loads of pathogenic bacteria in the blood using ddPCR at different time points until the last blood sample is taken on day 28-30 or the patient is discharged from the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Patients with first diagnosis of sepsis after ICU admission

Exclusion Criteria:

* Age under 18 years
* Do not meet Sepsis 3.0 diagnostic criteria
* Refusal to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to ICU
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Nucleic acid load of pathogenic bacteria at different time points | ''Nucleic acid load of pathogenic bacteria in the blood versus time'' could have a time frame of ''0, 2-3, 4-5, 6-7, 8-9, 10-12, 13-15, 20-22, 28-30 days post admission to the ICU with the first diagnosis of sepsis''.

SECONDARY OUTCOMES:
28-day mortality | Survival status at 28 days after the first diagnosis of sepsis on admission to the ICU

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Critical Care Medicine, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, China

IPD SHARING:
Plan to Share IPD: No